CLINICAL TRIAL: NCT05317715
Title: "Evaluation of the Impact of an Oral and Practical Presentation of Intrauterine Devices by a Health Professional on Women's Opinion as a Possible Contraceptive Method"
Brief Title: Evaluation of the Impact of an Oral and Practical Presentation of Intrauterine Devices by a Health Professional on Women's Opinion as a Possible Contraceptive Method
Acronym: EPODIU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Raincy Montfermeil Hospital Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GHT-GHI LRM-20220118
Record Dates: First submitted 2022-03-21; First posted 2022-04-08 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-03

CONDITIONS: Acceptance Processes
Keywords: Contraception; Intrauterine devices
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Single-centre, prospective, randomised, open-label study comparing a group of patients who had information and demonstration about IUDs prior to completing a questionnaire and a group of patients who did not have information and demonstration about IUDs prior to completing the questionnaire
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- without device information (Other): this group of patients will complete a questionnaire before receiving information on contraceptive intrauterine devices (copper or hormonal)
  Interventions: Other: Group A, who will complete a questionnaire before receiving information about intrauterine devices
- with device information (Other): This group of patients will receive information about contraceptive intrauterine devices (copper or hormonal) before completing a questionnaire
  Interventions: Other: Group B who will answer a questionnaire after having the information about the intrauterine devices

INTERVENTIONS:
Other: Group A, who will complete a questionnaire before receiving information about intrauterine devices — Group A will complete a questionnaire before receiving information about intrauterine devices and a demonstration of insertion/removal on a plastic dummy uterus.
  Arms: without device information
Other: Group B who will answer a questionnaire after having the information about the intrauterine devices — Group B will complete a questionnaire after receiving information about IUDs and a demonstration of insertion/removal on a plastic dummy uterus.
  Arms: with device information

SUMMARY:
Contraception among women in France has evolved considerably and has become a frequent reason for consultation in general practice in view of the growing shortage of gynaecologists practising in towns.

Intrauterine devices (IUDs) are the leading reversible contraceptive method used in the world, but only 20.7% of women in France were using them in 2010.

In practice, in France, use of the IUD is still "reserved" for older women or those who have already had children, despite medical recommendations.

In this study the investigator will investigate whether clear information about the mode of action and insertion/withdrawal of IUDs would dispel these misconceptions of patients.

DETAILED DESCRIPTION:
Contraception among women in France has evolved considerably and has become a frequent reason for consultation in general practice in view of the growing shortage of gynaecologists practising in towns.

Intrauterine devices (IUDs) are the leading reversible contraceptive method used in the world, but only 20.7% of women in France were using them in 2010.

In practice in France, the use of IUDs is still "reserved" for older women or those who have already had children, despite medical recommendations. Indeed, there is a certain feeling of mistrust towards the IUD as a contraceptive method. Sometimes the patient's reasons for refusal were unclear or misconceptions and prejudices prevailed.

Various research studies and theses have identified the various obstacles to the use of the IUD as a contraceptive. Today it would be interesting to evaluate whether a short presentation of the IUD during a consultation would lead to a better acceptance of women to use it as a possible contraceptive method.

In this study the investigators will investigate whether clear information about the mode of action and insertion/removal of IUDs would dispel these misconceptions of patients.

ELIGIBILITY:
Inclusion Criteria:

* Any woman aged 18 years and over who comes to a family planning centre
* Having expressed her free and informed written consent
* Affiliated to a social security scheme

Exclusion Criteria:

* Women under 18 years of age
* Woman with an IUD
* Woman who has had an IUD before
* Woman whose reason for consultation of the day is the insertion of an IUD
* Menopausal woman
* Woman who is infertile for any reason
* Illiterate woman or woman who does not read French
* Refusal to participate in the protocol
* Incapable of age.
* Pregnant or breastfeeding women
* Vulnerable persons and protected persons as provided for in the Public Health Code Public Health Code (articles L. 1121-5 to L.1121-8 and L.1122-1-2).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2022-08-14 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Rate of acceptance of the IUD as a possible contraceptive method | day 1
  measuring the acceptance rate of the intrauterine device as a potential contraceptive method

SECONDARY OUTCOMES:
Basic knowledge of intrauterine devices | day 1
  verification of Basic knowledge of intrauterine devices

CONTACTS AND LOCATIONS:
Overall Officials: Jean GUILLEMINOT, MD, Principal Investigator — Le Raincy Montfermeil hospital
Locations (1):
- Le Raincy Montfermeil hospital, Montfermeil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The delivery of information by the health professional to the patient about contraception: a descriptive cross-sectional study — https://dumas.ccsd.cnrs.fr/dumas-02883692/document